CLINICAL TRIAL: NCT03200587
Title: A Phase 1B, Open Label, Dose-finding Study to Evaluate the Safety and Tolerability of Cabometyx and Avelumab in Patients With Metastatic Renal Cell Carcinoma (mRCC)
Brief Title: Cabometyx and Avelumab in Patients With Metastatic Renal Cell Carcinoma (mRCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI102309
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — avelumab; cabozantinib

STUDY DESIGN:
Intervention Model Description: A phase 1B, open label, dose-finding study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab and cabozantinib, all patients (Experimental)
  Interventions: Drug: Avelumab; Drug: Cabozantinib

INTERVENTIONS:
Drug: Avelumab — Avelumab 10 mg/kg infusion every 2 weeks (Days 1 and 15) of every 28 day cycle for up to 12 cycles
Drug: Cabozantinib — Cabozantinib oral daily at 20 (starting dose 1), 40 (Dose Level 2) or 60 mg (Dose Level 3)
  Other Names: Cabometyx

SUMMARY:
This is an open-label, non-controlled, non-randomized, phase I dose-finding, of Cabometyx + Avelumab, to establish safety, feasibility, and the maximum tolerated dose (MTD) or Recommended Phase 2 Dose (RP2D) of Cabometyx in combination with Avelumab, and to investigate preliminary efficacy. The MTD or RP2D determined in this study will be used for a future study to formally test efficacy. The MTD determined by dose escalation will be the recommended Phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

Optional Pre-Screening Eligibility for Patients Scheduled for Cytoreductive Nephrectomy

* Male or female subject aged ≥ 18 years.
* Clinically, subject is a candidate for RCC diagnostic procedure (biopsy or surgery).
* Subject meets standard of care eligibility criteria for consideration of treatment with immunotherapy using a checkpoint inhibitor following surgical resection or biopsy.

Treatment Inclusion

* Male or female subject aged ≥ 18 years.
* Histologically proven renal cell carcinoma with a clear cell component.
* Radiographic evidence of metastatic disease.
* Measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) Score 0-2
* Adequate organ function as described in the protocol
* Negative serum or urine pregnancy test at screening for women of childbearing potential
* Highly effective contraception for both male and female subjects throughout the study and for at least 120 days after last Avelumab treatment administration if the risk of conception exists
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Current use of immunosuppressive medication, EXCEPT for the following:

  1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
  2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
  3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent per treating physician's clinical judgment. Subjects with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Active infection requiring intravenous antibiotics (antibiotics should have been completed prior to registration).
* Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. If the patient has a history of HBV or HCV then confirmatory polymerase chain reaction (PCR) testing is required to confirm the disease is not active.
* Live vaccinations within 4 weeks of the first dose of Avelumab and while on trial is prohibited.
* Prior exposure to checkpoint therapy or Cabozantinib.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Subjects taking prohibited medications as described in protocol. A washout period of prohibited medications for a period of at least two weeks or as clinically indicated should occur prior to the start of treatment
* Pregnant women or lactating women who are breastfeeding are excluded from this study.
* Stroke (including transient ischemic attack (TIA), myocardial infarction, or other ischemic event or symptomatic pulmonary embolism (PE) less than or equal to 6 months before dose of Cabometyx.
* Subjects with a diagnosis of deep vein thrombosis (DVT) or incidentally detected asymptomatic PE on routine scans are allowed if stable and treated with therapeutic anticoagulation for at least 2 weeks before first dose.
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Determine the recommended Phase II dose | 1 cycle (28 days)
  To assess the safety and tolerability of Avelumab + Cabometyx in subjects with mRCC and determine the recommended Phase II dose (RP2D). Safety, tolerability, adverse events (AEs), serious adverse events (SAEs), dose-limiting toxicities (DLTs).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2 years (Most patients are expected to be on treatment for approximately 10 months)
  To describe the clinical activity of Avelumab + Cabometyx in subjects with mRCC

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Agarwal, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Sahu KK, Brundage J, Benson M, Swami U, Boucher KM, Gupta S, Hawks J, Sirohi D, Agarwal N, Maughan BL. Phase I Trial of Combination Therapy With Avelumab and Cabozantinib in Patients With Newly Diagnosed Metastatic Clear Cell Renal Cell Carcinoma. Oncologist. 2023 Aug 3;28(8):737-e693. doi: 10.1093/oncolo/oyad019. PMID 36952231